CLINICAL TRIAL: NCT01427712
Title: Special Investigation (All Cases) of LipaCreon in Patients With Pancreatic Exocrine Insufficiency Due to Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Mylan Inc. (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Other Study IDs: P12-893
Record Dates: First submitted 2011-08-31; First posted 2011-09-02 (Estimated); Results first posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-03

CONDITIONS: Cystic Fibrosis; Exocrine Pancreatic Insufficiency; Pancreatic Diseases; Digestive System Diseases
Keywords: Digestive System Diseases; Cystic Fibrosis; Therapeutic Uses; Gastrointestinal Agents; Pancreatic Diseases; Pancrelipase; Exocrine Pancreatic Insufficiency
MeSH Terms: conditions — Cystic Fibrosis; Exocrine Pancreatic Insufficiency; Pancreatic Diseases; Digestive System Diseases | interventions — Pancrelipase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- LipaCreon: In general, pancrelipase 600 mg/dose was orally administered immediately after a meal, 3 times a day.
  Also, the dose was adjusted appropriately according to the patient's condition.
  Interventions: Drug: Pancrelipase

INTERVENTIONS:
Drug: Pancrelipase
  Other Names: Lipacreon

SUMMARY:
This study aims at collecting the information related to the safety and effectiveness in the pancreatic exocrine insufficiency patients due to cystic fibrosis receiving the treatment with LipaCreon in order to evaluate the effective and safe use of LipaCreon.

ELIGIBILITY:
Inclusion Criteria

* Patients who receive LipaCreon for the replacement of pancreatic digestive enzymes in pancreatic exocrine insufficiency due to cystic fibrosis

Exclusion Criteria

* Patients with a history of hypersensitivity to the ingredient of LipaCreon.
* Patients with a history of hypersensitivity to porcine protein

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who receive LipaCreon for the replacement of pancreatic digestive enzymes in pancreatic exocrine insufficiency
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shigenori Haruna, Study Director — Mylan EPD G.K.
Locations (21):
- Japan (21):
  - Site Reference ID/Investigator# 73813, Aichi
  - Site reference ID/Investigator # 96698, Aichi
  - Research facility ID ORG-000141, Aichi
  - Site reference ID/Investigator no. ORG-000842, Aichi
  - Site reference ID/Investigator # 93736, Aichi
  - Research facility ORG-000972, Ehime
  - Mylan investigational site A, Hyōgo
  - Site reference ID/Investigator # 93735, Ibaraki
  - Site Reference ID/Investigator# 88673, Ibaraki
  - Site Reference ID/Investigator# 65529, Ishikawa
  - Site Reference ID/Investigator# 65530, Kagawa
  - Site Reference ID/Investigator# 65527, Kagoshima
  - Mylan investigational site C, Kanagawa
  - Site Reference ID/Investigator# 65528, Miyagi
  - Mylan investigational site B, Miyagi
  - Research facility ID ORG-000594, Osaka
  - Research facility ID ORG-001138, Ōita
  - Research facility ORG-000971, Shizuoka
  - Site reference ID/Investigator# 117495, Tochigi
  - Research facility no. ORG-001309, Tokyo
  - Site Reference ID/Investigator# 67122, Tokyo

IPD SHARING:
Plan to Share IPD: Undecided
We will consider after completion of CSR

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For this survey, the contract for the conduct of the survey was concluded with 21 departments of 21 facilities during the period from August 2011 to March 2018. Among these, 24 patients were registered at 21 departments of 21 facilities (patient registration period: August 2011 to March 2017).
Groups:
- LipaCreon: In general, pancrelipase 600 mg/dose was orally administered immediately after a meal, 3 times a day.
  Also, the dose was adjusted appropriately according to the patient's condition.
  Pancrelipase
Period: Overall Study
Arm/Group | LipaCreon
Started | 24
Collected CRFs | 21
Safety Analysis Set | 21
Completed | 17
Not Completed | 7
Not completed — Transfer to a different hospital | 2
Not completed — Lost to Follow-up | 1
Not completed — Aggravation of cystic fibrosis | 3
Not completed — Failure to visit | 1

BASELINE CHARACTERISTICS:
Population: 21 are effective number for safety analysis.
Arm/Group | LipaCreon
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.7 (9.4)
Age, Customized [Count of Participants; unit: Participants]
  < 6 years | 12
  >= 6 years and < 12 years | 4
  >= 12 years and < 18 years | 0
  >= 18 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 21
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Japan | 21
Body Mass Index (BMI) [Count of Participants; unit: Participants]
  < 18.5 kg/m^2 | 16
  >= 18.5 kg/m^2 and < 25 kg/m^2 | 2
  >= 25 kg/m^2 | 0
  unknown | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Drug Reaction
Description: An adverse event (AE) was defined as any unfavourable or unintended disease, or symptom or sign of such a disease, or abnormal laboratory finding that occurred in a patient who received Lipacreon, whether or not considered related to the medicinal product. Also, an AE for which the relationship with Lipacreon could not be ruled out was regarded as an adverse drug reaction (ADR).
  1. Related : There is a temporal relationship between the use of the medicinal product and the onset of an AE, or a relapse with readministration,where other factors are less likely to be involved.
  2. Relationship cannot be ruled out : There are other potential factors although there is a temporal relationship between the use of the medicinal product and the onset of an AE
Time Frame: From the start of Lipacreon treatment to the end of the observation period or discontinuation. Approximately 7 years in the study completers (From date of dosage start, up to 7 years).
Population: Among the 21 patients from whom the survey forms were collected, no patient was excluded from the safety analysis or efficacy analysis, and both the safety analysis set and the efficacy analysis set included 21 patients.
Measure: Number; unit: participants
Arm/Group | LipaCreon
Number analyzed (Participants) | 21
participants | 1

2. Secondary Outcome: Nutritional Endpoints - BMI
Description: The following nutritional endpoints were measured prior to the start of Lipacreon treatment, at 4, 8, and 24 weeks after the start of treatment, at the completion of the 52-week observation period, at 1-year intervals during the follow-up period, and at the completion of follow-up in March 2018.
  •BMI (height [only prior to the start of Lipacreon treatment] and weight)
Time Frame: Baseline, 4 weeks, 8 weeks, 24 weeks, 52 weeks, 2 years, 3 years, 4 years, 5 years, 6 years, and 7 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | LipaCreon
Number analyzed (Participants) | 21
kg/m^2
  Baseline: number analyzed (Participants) | 18
  Baseline | 15.093 (1.955)
  4 weeks: number analyzed (Participants) | 12
  4 weeks | 15.583 (1.511)
  8 weeks: number analyzed (Participants) | 8
  8 weeks | 15.649 (1.667)
  24 weeks: number analyzed (Participants) | 13
  24 weeks | 15.604 (1.350)
  52 weeks: number analyzed (Participants) | 7
  52 weeks | 15.698 (1.239)
  2 years: number analyzed (Participants) | 9
  2 years | 15.766 (1.438)
  3 years: number analyzed (Participants) | 8
  3 years | 15.152 (1.241)
  4 years: number analyzed (Participants) | 6
  4 years | 15.479 (1.757)
  5 years: number analyzed (Participants) | 5
  5 years | 15.584 (2.608)
  6 years: number analyzed (Participants) | 4
  6 years | 15.819 (2.467)
  7 years: number analyzed (Participants) | 1
  7 years | 11.806

3. Secondary Outcome: Nutritional Endpoints - Serum Total Protein
Description: The following nutritional endpoints were measured prior to the start of Lipacreon treatment, at 4, 8, and 24 weeks after the start of treatment, at the completion of the 52-week observation period, at 1-year intervals during the follow-up period, and at the completion of follow-up in March 2018.
  •Serum total protein
Time Frame: Baseline, 4 weeks, 8 weeks, 24 weeks, 52 weeks, 2 years, 3 years, 4 years, 5 years, 6 years, and 7 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | LipaCreon
Number analyzed (Participants) | 21
g/dL
  Baseline: number analyzed (Participants) | 19
  Baseline | 7.282 (1.105)
  4 weeks: number analyzed (Participants) | 12
  4 weeks | 6.925 (0.770)
  8 weeks: number analyzed (Participants) | 8
  8 weeks | 6.700 (0.441)
  24 weeks: number analyzed (Participants) | 10
  24 weeks | 7.350 (1.049)
  52 weeks: number analyzed (Participants) | 8
  52 weeks | 7.421 (0.877)
  2 years: number analyzed (Participants) | 7
  2 years | 7.563 (1.058)
  3 years: number analyzed (Participants) | 7
  3 years | 8.029 (1.164)
  4 years: number analyzed (Participants) | 6
  4 years | 8.127 (1.301)
  5 years: number analyzed (Participants) | 4
  5 years | 7.390 (1.086)
  6 years: number analyzed (Participants) | 3
  6 years | 7.200 (0.557)
  7 years: number analyzed (Participants) | 1
  7 years | 6.100

4. Secondary Outcome: Nutrition Endpoints - Albumin
Description: The following nutritional endpoints were measured prior to the start of Lipacreon treatment, at 4, 8, and 24 weeks after the start of treatment, at the completion of the 52-week observation period, at 1-year intervals during the follow-up period, and at the completion of follow-up in March 2018.
  •Albumin
Time Frame: Baseline, 4 weeks, 8 weeks, 24 weeks, 52 weeks, 2 years, 3 years, 4 years, 5 years, 6 years, and 7 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | LipaCreon
Number analyzed (Participants) | 21
g/dL
  Baseline: number analyzed (Participants) | 19
  Baseline | 3.872 (0.641)
  4 weeks: number analyzed (Participants) | 13
  4 weeks | 4.054 (0.657)
  8 weeks: number analyzed (Participants) | 9
  8 weeks | 4.067 (0.339)
  24 weeks: number analyzed (Participants) | 10
  24 weeks | 4.130 (0.267)
  52 weeks: number analyzed (Participants) | 10
  52 weeks | 4.232 (0.549)
  2 years: number analyzed (Participants) | 8
  2 years | 4.390 (0.304)
  3 years: number analyzed (Participants) | 7
  3 years | 4.054 (0.323)
  4 years: number analyzed (Participants) | 5
  4 years | 4.040 (0.844)
  5 years: number analyzed (Participants) | 3
  5 years | 3.613 (0.931)
  6 years: number analyzed (Participants) | 3
  6 years | 4.233 (0.115)
  7 years: number analyzed (Participants) | 1
  7 years | 3.700

5. Secondary Outcome: Nutrition Endpoints - Total Cholesterol
Description: The following nutritional endpoints were measured prior to the start of Lipacreon treatment, at 4, 8, and 24 weeks after the start of treatment, at the completion of the 52-week observation period, at 1-year intervals during the follow-up period, and at the completion of follow-up in March 2018.
  •Total cholesterol
Time Frame: Baseline, 4 weeks, 8 weeks, 24 weeks, 52 weeks, 2 years, 3 years, 4 years, 5 years, 6 years, and 7 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | LipaCreon
Number analyzed (Participants) | 21
mg/dL
  Baseline: number analyzed (Participants) | 17
  Baseline | 124.94 (31.04)
  4 weeks: number analyzed (Participants) | 10
  4 weeks | 126.10 (34.94)
  8 weeks: number analyzed (Participants) | 6
  8 weeks | 128.00 (35.96)
  24 weeks: number analyzed (Participants) | 8
  24 weeks | 139.13 (40.88)
  52 weeks: number analyzed (Participants) | 9
  52 weeks | 123.11 (29.40)
  2 years: number analyzed (Participants) | 6
  2 years | 148.17 (26.12)
  3 years: number analyzed (Participants) | 6
  3 years | 139.00 (39.72)
  4 years: number analyzed (Participants) | 4
  4 years | 136.50 (30.88)
  5 years: number analyzed (Participants) | 2
  5 years | 114.00 (62.23)
  6 years: number analyzed (Participants) | 2
  6 years | 157.50 (57.28)
  7 years: number analyzed (Participants) | 1
  7 years | 167.00

6. Secondary Outcome: Nutrition Endpoints - Triglycerides
Description: The following nutritional endpoints were measured prior to the start of Lipacreon treatment, at 4, 8, and 24 weeks after the start of treatment, at the completion of the 52-week observation period, at 1-year intervals during the follow-up period, and at the completion of follow-up in March 2018.
  •Triglycerides
Time Frame: Baseline, 4 weeks, 8 weeks, 24 weeks, 52 weeks, 2 years, 3 years, 4 years, 5 years, 6 years, and 7 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | LipaCreon
Number analyzed (Participants) | 21
mg/dL
  Baseline: number analyzed (Participants) | 15
  Baseline | 81.6 (41.4)
  4 weeks: number analyzed (Participants) | 10
  4 weeks | 126.1 (115.2)
  8 weeks: number analyzed (Participants) | 6
  8 weeks | 73.2 (35.4)
  24 weeks: number analyzed (Participants) | 8
  24 weeks | 80.5 (39.6)
  52 weeks: number analyzed (Participants) | 7
  52 weeks | 117.1 (51.1)
  2 years: number analyzed (Participants) | 5
  2 years | 83.6 (69.9)
  3 years: number analyzed (Participants) | 4
  3 years | 89.8 (34.8)
  4 years: number analyzed (Participants) | 3
  4 years | 100.0 (49.2)
  5 years: number analyzed (Participants) | 2
  5 years | 89.0 (28.3)
  6 years: number analyzed (Participants) | 2
  6 years | 124.5 (38.9)
  7 years: number analyzed (Participants) | 1
  7 years | 160.0

7. Secondary Outcome: Nutrition Endpoints - Haemoglobin
Description: The following nutritional endpoints were measured prior to the start of Lipacreon treatment, at 4, 8, and 24 weeks after the start of treatment, at the completion of the 52-week observation period, at 1-year intervals during the follow-up period, and at the completion of follow-up in March 2018.
  •Haemoglobin
Time Frame: Baseline, 4 weeks, 8 weeks, 24 weeks, 52 weeks, 2 years, 3 years, 4 years, 5 years, 6 years, and 7 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | LipaCreon
Number analyzed (Participants) | 21
g/dL
  Baseline: number analyzed (Participants) | 19
  Baseline | 12.02 (1.84)
  4 weeks: number analyzed (Participants) | 13
  4 weeks | 12.38 (1.65)
  8 weeks: number analyzed (Participants) | 9
  8 weeks | 12.07 (1.94)
  24 weeks: number analyzed (Participants) | 11
  24 weeks | 12.82 (1.65)
  52 weeks: number analyzed (Participants) | 10
  52 weeks | 12.89 (1.88)
  2 years: number analyzed (Participants) | 8
  2 years | 13.41 (1.18)
  3 years: number analyzed (Participants) | 6
  3 years | 13.18 (0.81)
  4 years: number analyzed (Participants) | 5
  4 years | 13.38 (2.25)
  5 years: number analyzed (Participants) | 4
  5 years | 11.65 (2.11)
  6 years: number analyzed (Participants) | 3
  6 years | 12.50 (3.22)
  7 years: number analyzed (Participants) | 1
  7 years | 12.20

8. Secondary Outcome: Symptoms Related to Exocrine Pancreatic Insufficiency - Steatorrhoea
Description: The following symptoms were assessed as those related to exocrine pancreatic insufficiency prior to the start of Lipacreon treatment, at 4, 8, and 24 weeks after the start of treatment, at the completion of the 52-week observation period, at 1-year intervals during the follow-up period, and at the completion of follow-up in March 2018.
  •Steatorrhoea (Yes/No)
Time Frame: Baseline, 4 weeks, 8 weeks, 24 weeks, 52 weeks, 2 years, 3 years, 4 years, 5 years, 6 years, and 7 years
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | LipaCreon
Number analyzed (Participants) | 21
participants
  Baseline, Yes: number analyzed (Participants) | 18
  Baseline, Yes | 14
  Baseline, No: number analyzed (Participants) | 18
  Baseline, No | 4
  4 weeks, Yes: number analyzed (Participants) | 12
  4 weeks, Yes | 4
  4 weeks, No: number analyzed (Participants) | 12
  4 weeks, No | 8
  8 weeks, Yes: number analyzed (Participants) | 9
  8 weeks, Yes | 2
  8 weeks, No: number analyzed (Participants) | 9
  8 weeks, No | 7
  24 weeks, Yes: number analyzed (Participants) | 14
  24 weeks, Yes | 4
  24 weeks, No: number analyzed (Participants) | 14
  24 weeks, No | 10
  52 weeks, Yes: number analyzed (Participants) | 12
  52 weeks, Yes | 3
  52 weeks, No: number analyzed (Participants) | 12
  52 weeks, No | 9
  2 years, Yes: number analyzed (Participants) | 10
  2 years, Yes | 3
  2 years, No: number analyzed (Participants) | 10
  2 years, No | 7
  3 years, Yes: number analyzed (Participants) | 8
  3 years, Yes | 2
  3 Years, No: number analyzed (Participants) | 8
  3 Years, No | 6
  4 years, Yes: number analyzed (Participants) | 8
  4 years, Yes | 2
  4 years, No: number analyzed (Participants) | 8
  4 years, No | 6
  5 years, Yes: number analyzed (Participants) | 6
  5 years, Yes | 2
  5 years, No: number analyzed (Participants) | 6
  5 years, No | 4
  6 years, Yes: number analyzed (Participants) | 4
  6 years, Yes | 2
  6 years, No: number analyzed (Participants) | 4
  6 years, No | 2
  7 years, Yes: number analyzed (Participants) | 1
  7 years, Yes | 0
  7 years, No: number analyzed (Participants) | 1
  7 years, No | 1

9. Secondary Outcome: Symptoms Related to Exocrine Pancreatic Insufficiency - Frequency of Bowel Movements
Description: The following symptoms were assessed as those related to exocrine pancreatic insufficiency prior to the start of Lipacreon treatment, at 4, 8, and 24 weeks after the start of treatment, at the completion of the 52-week observation period, at 1-year intervals during the follow-up period, and at the completion of follow-up in March 2018.
  •Frequency of bowel movements (times/day)
Time Frame: Baseline, 4 weeks, 8 weeks, 24 weeks, 52 weeks, 2 years, 3 years, 4 years, 5 years, 6 years, and 7 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: times/day
Arm/Group | LipaCreon
Number analyzed (Participants) | 21
times/day
  Baseline: number analyzed (Participants) | 15
  Baseline | 2.40 (1.76)
  4 weeks: number analyzed (Participants) | 10
  4 weeks | 1.90 (0.74)
  8 weeks: number analyzed (Participants) | 7
  8 weeks | 1.86 (0.69)
  24 weeks: number analyzed (Participants) | 12
  24 weeks | 1.83 (0.83)
  52 weeks: number analyzed (Participants) | 11
  52 weeks | 1.82 (0.75)
  2 years: number analyzed (Participants) | 8
  2 years | 1.75 (1.16)
  3 years: number analyzed (Participants) | 8
  3 years | 1.63 (0.74)
  4 years: number analyzed (Participants) | 7
  4 years | 2.29 (1.11)
  5 years: number analyzed (Participants) | 5
  5 years | 1.60 (0.89)
  6 years: number analyzed (Participants) | 3
  6 years | 1.33 (0.58)
  7 years: number analyzed (Participants) | 1
  7 years | 1.00

10. Secondary Outcome: Symptoms Related to Exocrine Pancreatic Insufficiency - Diarrhoea
Description: The following symptoms were assessed as those related to exocrine pancreatic insufficiency prior to the start of Lipacreon treatment, at 4, 8, and 24 weeks after the start of treatment, at the completion of the 52-week observation period, at 1-year intervals during the follow-up period, and at the completion of follow-up in March 2018.
  •Diarrhoea (Yes/No)
Time Frame: Baseline, 4 weeks, 8 weeks, 24 weeks, 52 weeks, 2 years, 3 years, 4 years, 5 years, 6 years, and 7 years
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | LipaCreon
Number analyzed (Participants) | 21
participants
  Baseline, Yes: number analyzed (Participants) | 19
  Baseline, Yes | 6
  Baseline, No: number analyzed (Participants) | 19
  Baseline, No | 13
  4 weeks, Yes: number analyzed (Participants) | 13
  4 weeks, Yes | 1
  4 weeks, No: number analyzed (Participants) | 13
  4 weeks, No | 12
  8 weeks, Yes: number analyzed (Participants) | 10
  8 weeks, Yes | 0
  8 weeks, No: number analyzed (Participants) | 10
  8 weeks, No | 10
  24 weeks, Yes: number analyzed (Participants) | 16
  24 weeks, Yes | 0
  24 weeks, No: number analyzed (Participants) | 16
  24 weeks, No | 16
  52 weeks, Yes: number analyzed (Participants) | 13
  52 weeks, Yes | 1
  52 weeks, No: number analyzed (Participants) | 13
  52 weeks, No | 12
  2 years, Yes: number analyzed (Participants) | 11
  2 years, Yes | 1
  2 years, No: number analyzed (Participants) | 11
  2 years, No | 10
  3 years, Yes: number analyzed (Participants) | 8
  3 years, Yes | 1
  3 Years, No: number analyzed (Participants) | 8
  3 Years, No | 7
  4 years, Yes: number analyzed (Participants) | 9
  4 years, Yes | 0
  4 years, No: number analyzed (Participants) | 9
  4 years, No | 9
  5 years, Yes: number analyzed (Participants) | 7
  5 years, Yes | 0
  5 years, No: number analyzed (Participants) | 7
  5 years, No | 7
  6 years, Yes: number analyzed (Participants) | 4
  6 years, Yes | 0
  6 years, No: number analyzed (Participants) | 4
  6 years, No | 4
  7 years, Yes: number analyzed (Participants) | 1
  7 years, Yes | 0
  7 years, No: number analyzed (Participants) | 1
  7 years, No | 1

11. Secondary Outcome: Symptoms Related to Exocrine Pancreatic Insufficiency - Foul Stool Odour
Description: The following symptoms were assessed as those related to exocrine pancreatic insufficiency prior to the start of Lipacreon treatment, at 4, 8, and 24 weeks after the start of treatment, at the completion of the 52-week observation period, at 1-year intervals during the follow-up period, and at the completion of follow-up in March 2018.
  •Foul stool odour (Yes/No)
Time Frame: Baseline, 4 weeks, 8 weeks, 24 weeks, 52 weeks, 2 years, 3 years, 4 years, 5 years, 6 years, and 7 years
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | LipaCreon
Number analyzed (Participants) | 21
participants
  Baseline, Yes: number analyzed (Participants) | 19
  Baseline, Yes | 6
  Baseline, No: number analyzed (Participants) | 19
  Baseline, No | 13
  4 weeks, Yes: number analyzed (Participants) | 13
  4 weeks, Yes | 1
  4 weeks, No: number analyzed (Participants) | 13
  4 weeks, No | 12
  8 weeks, Yes: number analyzed (Participants) | 10
  8 weeks, Yes | 2
  8 weeks, No: number analyzed (Participants) | 10
  8 weeks, No | 8
  24 weeks, Yes: number analyzed (Participants) | 15
  24 weeks, Yes | 2
  24 weeks, No: number analyzed (Participants) | 15
  24 weeks, No | 13
  52 weeks, Yes: number analyzed (Participants) | 12
  52 weeks, Yes | 3
  52 weeks, No: number analyzed (Participants) | 12
  52 weeks, No | 9
  2 years, Yes: number analyzed (Participants) | 10
  2 years, Yes | 2
  2 years, No: number analyzed (Participants) | 10
  2 years, No | 8
  3 years, Yes: number analyzed (Participants) | 8
  3 years, Yes | 3
  3 Years, No: number analyzed (Participants) | 8
  3 Years, No | 5
  4 years, Yes: number analyzed (Participants) | 8
  4 years, Yes | 1
  4 years, No: number analyzed (Participants) | 8
  4 years, No | 7
  5 years, Yes: number analyzed (Participants) | 7
  5 years, Yes | 0
  5 years, No: number analyzed (Participants) | 7
  5 years, No | 7
  6 years, Yes: number analyzed (Participants) | 4
  6 years, Yes | 1
  6 years, No: number analyzed (Participants) | 4
  6 years, No | 3
  7 years, Yes: number analyzed (Participants) | 1
  7 years, Yes | 0
  7 years, No: number analyzed (Participants) | 1
  7 years, No | 1

12. Secondary Outcome: Symptoms Related to Exocrine Pancreatic Insufficiency - Inappetence
Description: The following symptoms were assessed as those related to exocrine pancreatic insufficiency prior to the start of Lipacreon treatment, at 4, 8, and 24 weeks after the start of treatment, at the completion of the 52-week observation period, at 1-year intervals during the follow-up period, and at the completion of follow-up in March 2018.
  •Inappetence (Yes/No)
Time Frame: Baseline, 4 weeks, 8 weeks, 24 weeks, 52 weeks, 2 years, 3 years, 4 years, 5 years, 6 years, and 7 years
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | LipaCreon
Number analyzed (Participants) | 21
participants
  Baseline, Yes: number analyzed (Participants) | 20
  Baseline, Yes | 7
  Baseline, No: number analyzed (Participants) | 20
  Baseline, No | 13
  4 weeks, Yes: number analyzed (Participants) | 13
  4 weeks, Yes | 0
  4 weeks, No: number analyzed (Participants) | 13
  4 weeks, No | 13
  8 weeks, Yes: number analyzed (Participants) | 10
  8 weeks, Yes | 0
  8 weeks, No: number analyzed (Participants) | 10
  8 weeks, No | 10
  24 weeks, Yes: number analyzed (Participants) | 16
  24 weeks, Yes | 4
  24 weeks, No: number analyzed (Participants) | 16
  24 weeks, No | 12
  52 weeks, Yes: number analyzed (Participants) | 13
  52 weeks, Yes | 2
  52 weeks, No: number analyzed (Participants) | 13
  52 weeks, No | 11
  2 years, Yes: number analyzed (Participants) | 11
  2 years, Yes | 3
  2 years, No: number analyzed (Participants) | 11
  2 years, No | 8
  3 years, Yes: number analyzed (Participants) | 8
  3 years, Yes | 2
  3 Years, No: number analyzed (Participants) | 8
  3 Years, No | 6
  4 years, Yes: number analyzed (Participants) | 9
  4 years, Yes | 3
  4 years, No: number analyzed (Participants) | 9
  4 years, No | 6
  5 years, Yes: number analyzed (Participants) | 7
  5 years, Yes | 3
  5 years, No: number analyzed (Participants) | 7
  5 years, No | 4
  6 years, Yes: number analyzed (Participants) | 4
  6 years, Yes | 1
  6 years, No: number analyzed (Participants) | 4
  6 years, No | 3
  7 years, Yes: number analyzed (Participants) | 1
  7 years, Yes | 0
  7 years, No: number analyzed (Participants) | 1
  7 years, No | 1

13. Secondary Outcome: Symptoms Related to Exocrine Pancreatic Insufficiency - Abdominal Distension
Description: The following symptoms were assessed as those related to exocrine pancreatic insufficiency prior to the start of Lipacreon treatment, at 4, 8, and 24 weeks after the start of treatment, at the completion of the 52-week observation period, at 1-year intervals during the follow-up period, and at the completion of follow-up in March 2018.
  •Abdominal distension (Yes/No)
Time Frame: Baseline, 4 weeks, 8 weeks, 24 weeks, 52 weeks, 2 years, 3 years, 4 years, 5 years, 6 years, and 7 years
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | LipaCreon
Number analyzed (Participants) | 21
participants
  Baseline, Yes: number analyzed (Participants) | 20
  Baseline, Yes | 5
  Baseline, No: number analyzed (Participants) | 20
  Baseline, No | 15
  4 weeks, Yes: number analyzed (Participants) | 13
  4 weeks, Yes | 1
  4 weeks, No: number analyzed (Participants) | 13
  4 weeks, No | 12
  8 weeks, Yes: number analyzed (Participants) | 10
  8 weeks, Yes | 2
  8 weeks, No: number analyzed (Participants) | 10
  8 weeks, No | 8
  24 weeks, Yes: number analyzed (Participants) | 16
  24 weeks, Yes | 2
  24 weeks, No: number analyzed (Participants) | 16
  24 weeks, No | 14
  52 weeks, Yes: number analyzed (Participants) | 13
  52 weeks, Yes | 1
  52 weeks, No: number analyzed (Participants) | 13
  52 weeks, No | 12
  2 years, Yes: number analyzed (Participants) | 11
  2 years, Yes | 3
  2 years, No: number analyzed (Participants) | 11
  2 years, No | 8
  3 years, Yes: number analyzed (Participants) | 8
  3 years, Yes | 0
  3 Years, No: number analyzed (Participants) | 8
  3 Years, No | 8
  4 years, Yes: number analyzed (Participants) | 9
  4 years, Yes | 1
  4 years, No: number analyzed (Participants) | 9
  4 years, No | 8
  5 years, Yes: number analyzed (Participants) | 7
  5 years, Yes | 3
  5 years, No: number analyzed (Participants) | 7
  5 years, No | 4
  6 years, Yes: number analyzed (Participants) | 4
  6 years, Yes | 0
  6 years, No: number analyzed (Participants) | 4
  6 years, No | 4
  7 years, Yes: number analyzed (Participants) | 1
  7 years, Yes | 0
  7 years, No: number analyzed (Participants) | 1
  7 years, No | 1

14. Secondary Outcome: Degree of General Improvement
Description: Degree of general improvement was assessed at 24 weeks after the start of Lipacreon treatment and at the completion of the 52-week observation period, using the following 4 grades:
  Improved, unchanged, exacerbated, unassessable
Time Frame: At 24 weeks
Population: Among the 21 patients from whom the survey forms were collected, no patient was excluded from the safety analysis or efficacy analysis, and both the safety analysis set and the efficacy analysis set included 21 patients. Of these 21 patients, 17 patients were obtained with data on Degree of General Improvement at 24 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | LipaCreon
Number analyzed (Participants) | 17
Participants
  Improved | 10
  Unchanged | 7
  Exacerbated | 0
  Unassessable | 0

15. Secondary Outcome: Degree of General Improvement
Description: as for outcome 14
Time Frame: At 52 weeks
Population: Among the 21 patients from whom the survey forms were collected, no patient was excluded from the safety analysis or efficacy analysis, and both the safety analysis set and the efficacy analysis set included 21 patients. Of these 21 patients, 14 patients were obtained with data on Degree of General Improvement at 52 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | LipaCreon
Number analyzed (Participants) | 14
Participants
  Improved | 9
  Unchanged | 5
  Exacerbated | 0
  Unassessable | 0

ADVERSE EVENTS:
Time Frame: From the start of Lipacreon treatment to the end of the observation period or discontinuation. Approximately 7 years in the study completers (From date of dosage start, up to 7 years).
Arm/Group | LipaCreon
All-Cause Mortality (participants affected / at risk) | 3/21
Serious Adverse Events (participants affected / at risk) | 4/21
Other Adverse Events (participants affected / at risk) | 4/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LipaCreon (N=21)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
C-Reactive Protein Increased (Investigations) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LipaCreon (N=21)
Bronchitis (Infections and infestations) | 2 (6)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2011-05-16): https://cdn.clinicaltrials.gov/large-docs/12/NCT01427712/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/12/NCT01427712/SAP_001.pdf